CLINICAL TRIAL: NCT05215418
Title: A Multicenter, Randomized, Double-Blind Study to Compare the Effects of VI-0521,Phentermine, and Placebo on Ambulatory Blood Pressure in Overweight or Obese Subjects
Brief Title: A Study of VI-0521 on Ambulatory Blood Pressure (ABPM) in Overweight or Obese Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OB-409
Record Dates: First submitted 2022-01-17; First posted 2022-01-31 (Actual); Results first posted 2024-06-18 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-06

CONDITIONS: Blood Pressure
Keywords: Obesity; Overweight; Qsymia; ABPM
MeSH Terms: conditions — Obesity; Overweight | interventions — Qsymia; Phentermine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) (Experimental): Week 1: VI-0521 (Phentermine 3.75 mg + Topiramate 23 mg) oral capsule, once daily; Week 2: VI-0521 (Phentermine 7.5 mg + Topiramate 46 mg) oral capsule, once daily; Week 3: VI-0521 (Phentermine 11.25 mg + Topiramate 69 mg) oral capsule, once daily; Weeks 4-8: VI-0521 (Phentermine 15 mg + Topiramate 92 mg) oral capsule, once daily
  Interventions: Drug: VI-0521
- Phentermine 30mg (Active Comparator): Weeks 1-8: Phentermine 30mg oral capsule, once daily
  Interventions: Drug: Phentermine
- Placebo (Placebo Comparator): Weeks 1-8: Placebo oral capsule, once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VI-0521 — Phentermine/Topiramate Top Dose 15 mg/92 mg capsule
  Other Names: Qsymia; Phentermine and topiramate
  Arms: VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg)
Drug: Phentermine — Phentermine 30 mg capsule
  Arms: Phentermine 30mg
Drug: Placebo — Inactive oral capsule
  Arms: Placebo

SUMMARY:
The study is being conducted to evaluate the effect of VI-0521 (Qsymia®) on blood pressure as measured by 24-hour ambulatory blood pressure monitoring, compared to both placebo and an active control (phentermine 30 mg).

ELIGIBILITY:
Inclusion Criteria:

* Overweight/obese adult males/females 18-75 years of age with a BMI ≥ 27 kg/m2;
* At least 1 weight-related comorbidity (i.e., hypertension, dyslipidemia, Type 2 diabetes mellitus [T2DM] or prediabetes, or obstructive sleep apnea).
* Must be ambulatory, willing, and able to wear ABPM monitor apparatus for 24 hours at beginning and end of study.

Exclusion Criteria:

* Screening blood pressure of > 140/90 mmHg;
* Type 1 diabetes; T2DM treated with SFUs, GLP-1 receptor agonists, SGLT inhibitors; or not on stable diabetic medications for at least 3 months prior to randomization;
* Clinically significant cardiac, hepatic, renal, pulmonary, or thyroid disease;
* History of bipolar disorder, psychosis, greater than one lifetime episode of major depressive disorder, or presence or history of suicidal behavior or suicidal ideation with intent to act;
* History of glaucoma;
* Night shift workers;
* Obesity of known genetic or endocrine origin; recent history of weight instability, or recent participation in a formal weight loss program within 3 months prior to screening; and
* Smoking cessation within 3 months prior to screening;
* Use of antihypertensive medications, antidiabetic medications, statins or other lipid lowering agents, or CPAP therapy that has not been stable for at least 3 months prior to randomization;
* COVID-19 vaccination or treatment for severe COVID-19 infection within a month prior to randomization.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 565 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-04-11 (Actual); Study Completion 2023-04-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Clinical Site, Anniston, Alabama
  - Clinical Site, Mobile, Alabama
  - Clinical Site, Lincoln, California
  - Clinical Site, Long Beach, California
  - Clinical Site, Sacramento, California
  - Clinical Site, Spring Valley, California
  - Clinical Site, Upland, California
  - Clinical Site, Washington D.C., District of Columbia
  - Clinical Site, Coral Gables, Florida
  - Clinical Site, Miami, Florida
  - Clinical Site, Port Orange, Florida
  - Clinical Site, Brownsburg, Indiana
  - Clinical Site, Evansville, Indiana
  - Clinical Site, Wichita, Kansas
  - Clinical Site, Lexington, Kentucky
  - Clinical Site, Louisville, Kentucky
  - Clinical Site, Baton Rouge, Louisiana
  - Clinical Site, Kansas City, Missouri
  - Clinical Site, Butte, Montana
  - Clinical Site, Cary, North Carolina
  - Clinical Site, Eugene, Oregon
  - Clinical Site, Columbia, South Carolina
  - Clinical Site, Knoxville, Tennessee
  - Clinical Site, Friendswood, Texas
  - Clinical Site, North Richland Hills, Texas
  - Clinical Site, San Antonio, Texas
  - Clinical site, Salt Lake City, Utah
  - Clinical Site, Norfolk, Virginia

REFERENCES:
- [Derived] Bays HE, Hsia DS, Nguyen LT, Peterson CA, Varghese ST. Effects of phentermine / topiramate extended-release, phentermine, and placebo on ambulatory blood pressure monitoring in adults with overweight or obesity: A randomized, multicenter, double-blind study. Obes Pillars. 2024 Jan 8;9:100099. doi: 10.1016/j.obpill.2024.100099. eCollection 2024 Mar. PMID 38304225

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) | Phentermine 30mg | Placebo
Started | 190 | 191 | 184
Completed | 156 | 167 | 164
Not Completed | 34 | 24 | 20

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) | Phentermine 30mg | Placebo | Total
Number analyzed (Participants) | 190 | 191 | 184 | 565
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (13.34) | 53.3 (12.12) | 53.3 (11.36) | 53.4 (12.29)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 142 | 137 | 415
  Male | 54 | 49 | 47 | 150
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 50 | 47 | 149
  Not Hispanic or Latino | 138 | 141 | 137 | 416
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 2 | 5
  Asian | 2 | 3 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 1 | 3
  Black or African American | 25 | 17 | 39 | 81
  White | 154 | 167 | 140 | 461
  More than one race | 2 | 0 | 2 | 4
  Unknown or Not Reported | 4 | 2 | 0 | 6
Region of Enrollment [Number; unit: participants]
  United States | 190 | 191 | 184 | 565
Hypertensive status [Count of Participants; unit: Participants]
  No Medical Diagnosis of or Treatment for Hypertension | 64 | 61 | 58 | 183
  Medical Diagnosis of Hypertension Treated with 0 to 2 Antihypertensive Agents | 116 | 120 | 117 | 353
  Medical Diagnosis of Hypertension Treated with 3 or More Antihypertensive Agents | 10 | 10 | 9 | 29
Diabetes Status [Count of Participants; unit: Participants]
  Type 2 Diabetes | 25 | 19 | 20 | 64
  Prediabetes | 27 | 24 | 25 | 76
  Gestational Diabetes | 1 | 0 | 0 | 1
  Borderline Diabetes | 0 | 0 | 1 | 1
  Not Diabetic | 137 | 148 | 138 | 423
Blood Pressure [Mean (Standard Deviation); unit: mmHg]
  Systolic Blood Pressure | 123.9 (9.82) | 123.4 (10.38) | 124.5 (11.23) | 123.9 (10.48)
  Diastolic Blood Pressure | 77.5 (7.63) | 77.0 (7.98) | 78.3 (7.71) | 77.6 (7.78)
Weight [Mean (Standard Deviation); unit: kg] | 98.8 (20.84) | 99.5 (21.58) | 100.4 (21.52) | 99.6 (21.29)
Height [Mean (Standard Deviation); unit: cm] | 165.7 (9.16) | 166.6 (9.51) | 166.1 (10.08) | 166.2 (9.58)
BMI (Body Mass Index) [Mean (Standard Deviation); unit: kg/m2] | 35.7 (6.20) | 35.4 (5.88) | 36.2 (6.17) | 35.8 (6.08)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 8 in Mean Systolic Blood Pressure as Measured by 24-hr ABPM
Description: The change between systolic blood pressure measured at Week 8 relative to the baseline measurements from the ABPM data read out. Blood pressure and heart rate were measured every 20 minutes from 6:00 to 22:00 hours, and every 30 minutes from 22:01 to 5:59 hours for 24 consecutive hours, while subjects continue normal routine activities.
Time Frame: Baseline to Week 8
Population: Subjects who completed the study per protocol. Per Protocol Population (PPP) was defined as:
  1. Randomized and received at least one dose of study drug;
  2. ≥ 80% treatment compliance;
  3. Last daily dose of study drug administered on the same date that ABPM was initiated at Week 8/End of Study or early termination (EOS);
  4. ≥ 23.5 hours of ABPM data at baseline and at Week 8/EOS or early termination, and ≥ 75% ABPM readings;
  5. No major protocol deviation that impacted ABPM readings.
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) | Phentermine 30mg | Placebo
Number analyzed (Participants) | 122 | 133 | 130
mmHg | -3.3 (1.07) | 1.4 (1.05) | -0.1 (1.04)
Statistical Analysis 1: Comparison: VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) vs Phentermine 30mg; Test type: Other — If the upper bound of the two-sided 95% confidence interval for the between-treatment group difference (VI-0521 minus placebo or phentermine) in change from baseline in 24-hr mean SBP was less than 3 mmHg, success for a non-inferiority test was claimed and the null hypothesis was rejected. If the upper bound of the two-sided 95% confidence interval was less than 0 mmHg, superiority was claimed; p < 0.001, ANCOVA
Statistical Analysis 2: Comparison: VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0059, ANCOVA
Statistical Analysis 3: Comparison: Phentermine 30mg vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.1867, ANCOVA

2. Secondary Outcome: Change From Baseline to Week 8 in Mean Diastolic Blood Pressure as Measured by 24-hr ABPM
Description: The change between diastolic blood pressure measured at Week 8 relative to the baseline measurements from the ABPM data read out. Blood pressure and heart rate were measured every 20 minutes from 6:00 to 22:00 hours, and every 30 minutes from 22:01 to 5:59 hours for 24 consecutive hours, while subjects continue normal routine activities.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) | Phentermine 30mg | Placebo
Number analyzed (Participants) | 122 | 133 | 130
mmHg | 0.8 (0.64) | 2.4 (0.64) | -0.4 (0.63)
Statistical Analysis 1: Comparison: VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) vs Phentermine 30mg; Test type: Other — If the upper bound of the two-sided 95% confidence interval for the between-treatment group difference (VI-0521 minus placebo or phentermine) in change from baseline in 24-hr mean DBP was less than 3 mmHg, success for a non-inferiority test was claimed and the null hypothesis was rejected. If the upper bound of the two-sided 95% confidence interval was less than 0 mmHg, superiority was claimed; p = 0.0277, ANCOVA
Statistical Analysis 2: Comparison: VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) vs Placebo; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0852, ANCOVA
Statistical Analysis 3: Comparison: Phentermine 30mg vs Placebo; Test type: Other — [test comment as in outcome 2, analysis 1]; p < .0001, ANCOVA

3. Secondary Outcome: Mean Change in Systolic and Diastolic Blood Pressure From Baseline to Week 8 as Measured in Clinic
Description: The change between systolic and diastolic blood pressure measured in the clinic at Week 8 relative to the baseline measurements after subjects are seated comfortably for at least 10 minutes prior to taking blood pressure. In clinic blood pressure for determining hypertension was the average of three successive blood pressure readings, collected at least 2 minutes apart. The mean of the three values was be recorded as the subject's blood pressure.
Time Frame: Baseline to Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mmHg
Arm/Group | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) | Phentermine 30mg | Placebo
Number analyzed (Participants) | 122 | 133 | 130
mmHg
  Systolic blood pressure as measured in clinic | -4.3 (1.15) | -1.2 (1.13) | -1.7 (1.12)
  Diastolic blood pressure as measured in clinic | -1.3 (0.82) | 1.0 (0.81) | -1.1 (0.80)
Statistical Analysis 1: Comparison: VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) vs Phentermine 30mg; In-clinic systolic blood pressure; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0109, ANCOVA
Statistical Analysis 2: Comparison: VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) vs Placebo; In-clinic systolic blood pressure; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.0339, ANCOVA
Statistical Analysis 3: Comparison: Phentermine 30mg vs Placebo; In-clinic systolic blood pressure; Test type: Other — [test comment as in outcome 1, analysis 1]; p = 0.6769, ANCOVA
Statistical Analysis 4: Comparison: VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) vs Phentermine 30mg; In-clinic diastolic blood pressure; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0082, ANCOVA
Statistical Analysis 5: Comparison: VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) vs Placebo; In-clinic diastolic blood pressure; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.8131, ANCOVA
Statistical Analysis 6: Comparison: Phentermine 30mg vs Placebo; In-clinic diastolic blood pressure; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.0150, ANCOVA

ADVERSE EVENTS:
Time Frame: Up to a total of 12 weeks (from baseline to 28 days after last dose of study drug)
Arm/Group | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) | Phentermine 30mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/190 | 0/191 | 0/184
Serious Adverse Events (participants affected / at risk) | 0/190 | 1/191 | 0/184
Other Adverse Events (participants affected / at risk) | 66/190 | 44/191 | 6/184
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) (N=190) | Phentermine 30mg (N=191) | Placebo (N=184)
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 — chest pain or discomfort due to coronary heart disease
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VI-0521 Top Dose (Phentermine 15 mg + Topiramate 92 mg) (N=190) | Phentermine 30mg (N=191) | Placebo (N=184)
Dry mouth (Gastrointestinal disorders) | 22 (22) | 22 (22) | 1 (1)
Constipation (Gastrointestinal disorders) | 7 (8) | 11 (11) | 2 (2)
Dizziness (Nervous system disorders) | 11 (13) | 9 (10) | 1 (1)
Paraesthesia (Nervous system disorders) | 18 (27) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (9) | 10 (10) | 1 (1)

LIMITATIONS AND CAVEATS:
Participants with baseline blood pressure greater than 140/90 were excluded. Of the 565 total participants randomized and treated with study drug, 180 participants were excluded from the per protocol population used for the primary analysis due to participants' reluctance or inability to properly complete end of study ABPM assessments.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/18/NCT05215418/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT05215418/SAP_001.pdf